CLINICAL TRIAL: NCT05202223
Title: Creating Harmony at HOME: A Pilot Study of a Telehealth Based Program for Rural Caregivers' Ability to Adapt Home Environments for Adults With ADRD
Brief Title: Harmony at Home: A Pilot Telehealth Program for Rural ADRD Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth K Rhodus (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Emory University (Other)
Responsible Party: Sponsor-Investigator, Elizabeth K Rhodus, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 66767; P30AG064200 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
Keywords: Telehealth; Caregiver burnout; Behavioral and psychological symptoms of dementia; BPSD; Environment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Caregiver Burden; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Harmony at HOME (Experimental): H@H is a 6-week telehealth intervention delivered by an occupational therapist during weekly visits.
  Interventions: Behavioral: Harmony at HOME (H@H)

INTERVENTIONS:
Behavioral: Harmony at HOME (H@H) — H@H is a 6-week telehealth intervention delivered by an occupational therapist during weekly visits.

SUMMARY:
There is a need for caregiver-initiated and -implemented non-pharmacological interventions directly to and for the person with dementia, including environmental assessment and modification, as first-line treatments for behavioral and psychological symptoms of dementia (BPSD) in persons living with dementia (PLWD). Delivered via telehealth, Harmony at HOME (H@H) aims to train caregivers of persons with moderate to severe ADRD in the skills of assessing and modifying the home environment to promote "person-environment fit," a concept that posits that the ability to access features within a built environment (e.g. bathroom, stairs,) or that factors within the environment itself (lighting, noise level, temperature), especially when linked with individualized social support, contribute to or even shape behavior.

In addition to the intervention, the first 10 caregiver participants to enroll will also be invited to participate in two focus groups that will be facilitated during and after the intervention. The first focus group focuses on experiences as a dementia caregiver in rural areas. The second focus group focuses on providing feedback regarding caregivers' perceptions, acceptability, and usefulness of the H@H intervention. These focus groups will be conducted as structured interviews with open-ended questions that encourage participants to share their experiences.

DETAILED DESCRIPTION:
Behavioral disruptions by individuals with Alzheimer's disease and related dementias (ADRD) are reported in nearly 90% of persons living with ADRD. Such behavioral and psychological symptoms of dementia (BPSD) are highly correlated with increased caregiver burden and burnout, decreased quality of life for the person living with dementia and their caregiver, institutionalization, and patient mortality. There is a need for caregiver-initiated and -implemented non-pharmacological interventions directly to and for the person with dementia, including environmental assessment and modification, as first-line treatments for BPSD in persons living with dementia (PLWD). Delivered via telehealth, Harmony at HOME (H@H) aims to train caregivers of persons with moderate to severe ADRD in the skills of assessing and modifying the home environment to promote "person-environment fit," a concept that posits that the ability to access features within a built environment (e.g. bathroom, stairs,) or that factors within the environment itself (lighting, noise level, temperature), especially when linked with individualized social support, contribute to or even shape behavior. In ideal circumstances, adults adjust or adapt to meet the demands of the environment; likewise, in the ideal, environments are designed in ways that facilitate positive behaviors. ADRD progressively interferes with an individual's capacity to self-optimize person-environment fit; in such cases, caregivers have the opportunity to create a supportive environment that negates some behavioral challenges and encourages functional activity engagement. H@H seeks to help caregivers acquire the skills and sense of mastery that will enable them to create such supportive environments within the homes of people with dementia. H@H will be tested with caregivers and the person living with dementia in the Appalachian region of rural Kentucky, a region with the poorest healthcare options for older adults in the country and plagued with extremely high rates of co-morbid conditions, including ADRD. Access to quality caregiver training, in-home caregiver support, and respite is significantly limited. This pilot study will enable the investigators not only to establish the feasibility of the program but to demonstrate this capacity with a population of caregivers and persons with dementia that is in particular need and difficult to reach.

ELIGIBILITY:
Inclusion and excluded groups: Recruitment and enrollment will be inclusive of all groups living within rural, Appalachia Kentucky who are over the age of 21.

Participants must meet all inclusion criteria in order to participate in the study:

Caregiver for Participant with Dementia:

1. Men or women aged 21-99, inclusive.
2. Willingness and ability to participate in trial and implement recommended intervention strategies throughout the duration of the study.
3. Access to and ability to use video technology (Zoom) for telehealth visits.
4. English speaking, able to read and write.
5. Ability to retrieve and return mail.

Participants with Dementia:

1. Men or women aged 65-99, inclusive.
2. Living at home in the community with one primary caregiver.
3. 3. Diagnosis of Alzheimer's disease as primary dementia type of moderate to severe stages (confirmed by Clinical Dementia Rating Scale score of 1.0+)
4. No change in medical condition for one month prior to screening visit
5. No change in medications for 4 weeks prior to screening visit.
6. If on psychotropic medication, the participant is at a point where dosage and treatment are stabilized for the duration of the study.
7. Physically acceptable for this study as confirmed by medical history, physical exam, and clinical tests completed by medical professional (MD, APRN, PA or OT).
8. Functional sensory abilities with or without aids (hearing, vision, smell, touch, taste)
9. Caregiver report of challenges related to behaviors within 4 weeks of study enrollment.
10. Caregiver willing to participant throughout duration of study.
11. Caregiver access to and ability to use video technology (Zoom, Skype, video call) which resembles telehealth visits.
12. Contact with University of Kentucky Alzheimer's Disease Center (UKADC) or Kentucky Neuroscience Institute (KNI) medical provider within 12 months of study recruitment.
13. Not actively participating in physical/occupational therapy throughout duration of study.

Exclusion Criteria

Caregiver for Participant with Dementia:

1. Diagnosis of mild cognitive impairment or dementia.
2. Severe psychological stress or active state of psychiatric conditions (severe depression, mania, hallucinations/delusions).

Participants with Dementia:

1. Unstable medical conditions within one month prior to screening visit such as poorly controlled blood pressure, diabetes, current cancer diagnosis, or breathing problems, etc.
2. Wheelchair or bed bound.
3. Residence in skilled nursing facility or facility-based care.
4. Skin lesions or skin abnormalities throughout upper extremities.
5. Allergies related to lotion or fragrance.
6. Caregiver report of physically violent behaviors.
7. Initiation of antipsychotic medication within 4 weeks prior to screening or unpredictable use of such medications
8. Diagnosis of profound or total sensory altering disorders including macular degeneration, legal blindness, total deafness, severe peripheral neuropathy, anosmia.
9. Major depression in past 12 months (DSM-IV criteria), major mental illness such as schizophrenia, bipolar disorder, personality disorders, or recent (in past 12 months) alcohol or substance abuse.
10. Diagnosis or concern of epilepsy.
11. Use of any investigational agents or devices within 30 days prior to screening.
12. Major infection within 4 weeks prior to the Baseline Visit.
13. Physically unacceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Jicha, MD, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhodus EK, Kryscio R, Jicha G, Baum C, Henley L, Fairchild V, Roberts C, Gibson A. Creating harmony at home via environmental cueing: A feasibility trial of a non-pharmacological intervention for rural caregivers of persons with dementia. Alzheimers Dement. 2025 Jul;21(7):e70405. doi: 10.1002/alz.70405. PMID 40621818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Harmony at HOME
Started | 80 (80 individuals were consented in dyads. 40 caregivers and 40 persons with cognitive impairment. 1 dyad dropped out prior to baseline data collection, therefore a total of 78 participants completed baseline data.)
Completed | 52 (26 dyads completed the intervention, this includes 26 caregivers and 26 individuals with cognitive impairment.)
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: 39 dyads completed baseline data collection (39 caregivers and 39 persons with cognitive impairment)
Arm/Group | Harmony at HOME
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only 78 participants completed baseline data collection
  years
    Caregiver: number analyzed (Participants) | 39
    Caregiver | 60.69 (1.99)
    Participant with Dementia: number analyzed (Participants) | 39
    Participant with Dementia | 78.74 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There was no response to this question for 8 participants
  Participants
    Caregiver: number analyzed (Participants) | 39
    Caregiver: Female | 6
    Caregiver: Male | 33
    Participant with Dementia: number analyzed (Participants) | 31
    Participant with Dementia: Female | 11
    Participant with Dementia: Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 78 completed baseline data collection
  Participants
    Caregiver: number analyzed (Participants) | 39
    Caregiver: Hispanic or Latino | 0
    Caregiver: Not Hispanic or Latino | 37
    Caregiver: Unknown or Not Reported | 2
    Participant with Dementia: number analyzed (Participants) | 39
    Participant with Dementia: Hispanic or Latino | 0
    Participant with Dementia: Not Hispanic or Latino | 29
    Participant with Dementia: Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 78 participants completed baseline data collection.
  Participants
    Caregiver: number analyzed (Participants) | 39
    Caregiver: American Indian or Alaska Native | 0
    Caregiver: Asian | 0
    Caregiver: Native Hawaiian or Other Pacific Islander | 0
    Caregiver: Black or African American | 1
    Caregiver: White | 35
    Caregiver: More than one race | 0
    Caregiver: Unknown or Not Reported | 3
    Participant with Dementia: number analyzed (Participants) | 39
    Participant with Dementia: American Indian or Alaska Native | 0
    Participant with Dementia: Asian | 0
    Participant with Dementia: Native Hawaiian or Other Pacific Islander | 0
    Participant with Dementia: Black or African American | 1
    Participant with Dementia: White | 30
    Participant with Dementia: More than one race | 0
    Participant with Dementia: Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Mastery
Description: Pearlin Mastery Scale: A 4-item scale measuring the extent to which a participant sees life as being under his/her personal control vs. something that is fatalistically ruled. Scores range from 4 to 16, with higher scores indicating greater levels of mastery.
Time Frame: baseline, visit 2 (week 6), visit 3 (week 10)
Population: Only caregiver data are reported for this outcome. 1 participant was unable to be contacted for visit 3 data collection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Harmony at HOME
Number analyzed (Participants) | 26
units on a scale
  Baseline | 12.6 (2.1)
  Visit 2 | 13 (1.6)
  Visit 3: number analyzed (Participants) | 25
  Visit 3 | 13 (1.7)

2. Other Pre Specified Outcome: Change in Caregiver Burden
Description: Zarit Burden Interview: It is a questionnaire consisting of 22 items. A minimum score of 0 and a maximum score of 88 can be obtained. The higher the scale score, the higher the difficulty experienced.
Time Frame: Timeframe 10 weeks (baseline, 6 weeks, 4 week follow up)]
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Caregiver Stress
Description: Perceived Stress Scale: Caregiver report of perceived stress. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent a worse outcome.
Time Frame: Timeframe 10 weeks (baseline, 6 weeks, 4 week follow up)]
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Caregiver Satisfaction
Description: Revised Caregiving Appraisal Scale, Sub-scale on caregiver satisfaction: Care partner satisfaction consisting of 6-items, 5-point Likert scale. Higher score indicates greater satisfaction.
Time Frame: Timeframe 10 weeks (baseline, 6 weeks, 4 week follow up)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Behavioral Symptoms of Person With Alzheimer's Disease
Description: Revised Memory and Behavior Problems Checklist: 24-item caregiver report measure, 5-point Likert scale, higher scores mean greater behavioral problems.
Time Frame: Timeframe 10 weeks (baseline, 6 weeks, 4 week follow up)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: All-Cause Mortality, Serious Adverse Events and Other Adverse Events were reported for participants with dementia. All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not monitored/assessed in caregiver participants.
Groups:
- Harmony at HOME: This is a single-arm study. Dyads (caregiver and person with dementia) were enrolled in the H@H telehealth intervention delivered by an occupational therapist during weekly visits.
  Participants were either 1) caregiver or 2) person with dementia (person at risk). Adverse Events are reported for persons with dementia.
Arm/Group | Harmony at HOME
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 14/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Harmony at HOME (N=40)
Fall (General disorders) | 12 — All AE reported were of the person with dementia (the person at risk).
Hospitalization (General disorders) | 2 — All AE reported were of the person with dementia (the person at risk).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT05202223/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT05202223/ICF_000.pdf